CLINICAL TRIAL: NCT03951376
Title: Universal Preventive Resilience Intervention Globally Implemented in Schools to Improve and Promote Mental Health for Teenagers
Brief Title: Universal Preventive Resilience Intervention to Improve and Promote Mental Health for Teenagers
Acronym: UPRIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosistemak Institute for Health Systems Research (Other)
Collaborators: Osakidetza (Other); Bruno Kessler Foundation (Unknown); Urzad Marszalkowski Wojewodztwa Dolnoslaskiego in Poland (Unknown); Norwegian University of Science and Technology (Other); Directorate of Health in Iceland (Unknown); University of Aarhus (Other); University of Iceland (Other); Daily Centre for Psychiatry and Speech Disorders Poland (Unknown); Falkiewicz Specialist Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 754919
Record Dates: First submitted 2019-05-08; First posted 2019-05-15 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Anxiety Symptoms; Depressive Symptoms; Behavioral Problem of Child; Mental Disorder in Adolescence; School Absenteeism; Bullying of Child; Cyberbullying; Violence in Adolescence
MeSH Terms: conditions — Anxiety Disorders; Depression; Cyberbullying

STUDY DESIGN:
Intervention Model Description: Cluster, randomized, controlled (two parallel groups) trial. The intervention is conducted in two phases (intensive phase and follow-up phase). The intervention is repeated 2 times during 3 years (2 waves)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The schools in this arm will implement the UPRIGHT programme (18 skills related to Mindfulness, Coping, Efficacy and Social and emotional learning) during a minimum of 18 sessions and a maximum of 24 in a period of 6 months, which will be conducted by teachers to adolescents of 1st grade (12-14 years of age).
  Teachers will be trained by the UPRIGHT team at the beginning of the school year (3 months) and families will have a combination of face to face training and online training throughout the UPRIGHT platform.
  Interventions: Behavioral: UPRIGHT intervention
- Control (No Intervention): Schools in the control arm have their usual curricula and are not provided of any intervention resources or support, apart from those in the common daily activities.

INTERVENTIONS:
Behavioral: UPRIGHT intervention — The UPRIGHT intervention design consists of two different phases consecutively implemented in two school years: intensive phase and follow-up phase. During the intensive phase, all stakeholders are trained in the UPRIGHT WELL-BEING FOR US programme (18 skills). The follow-up phase (WELL-BEING FOR ALL) intends not only to maintain the effect of the intensive training in youths, but also to boost the positive mental health atmosphere created in the whole school. To do so, different collective activities will be organized at school level such as celebration of thematic days, activities with the community, and outdoor/indoor activities.
  Arms: Intervention

SUMMARY:
Adolescence is a period of many physical, mental, emotional, and social changes. It is also associated with risk behaviour conducts. Nonetheless, not all youths under disadvantage, adversity, or exposure to risk factors experience negative mental health outcomes. The concept of RESILIENCE provides one possible explanation for the ability of some individuals to maintain positive mental health. Resilience is thus the ability of an individual or community to adapt to life challenges or adversities while maintaining mental health and well-being. The increasing prevalence of mental disorders amongst children (around 10-20% of young people) makes positive mental health promotion in schools necessary through intervention programmes. UPRIGHT (Universal Preventive Resilience Intervention Globally implemented in schools to improve and promote mental Health for Teenagers) is a research and innovation project funded by the European Union´s Horizon 2020 programme (No. 754919). UPRIGHT general aim is to promote mental well-being and prevent mental disorders in youth by enhancing resilience capacities. It has been designed as a whole school approach addressing early adolescents, their families and the school community to finally create a real mental well-being culture at schools.

DETAILED DESCRIPTION:
The operational objectives of UPRIGHT are:

* to co-create (involving adolescents, families, school staff, clinicians, policy makers) an innovative resilience holistic program in schools for the promotion of mental health in youth between 12 and 14 years;
* to deploy an intervention in five different pan-European regions;
* to better understand the natural history of mental disorders according to the resilience level and provide evidence of specific resilience factors promoting positive mental well-being longitudinally;
* to demonstrate the effectiveness and predict future impact of an intervention in terms of improvement of quality of life, mental well-being, and academic performance, and a reduction of absenteeism and bullying cases;
* to transfer the programme to Europe and beyond by disseminating the results and enabling innovative action plans for mental well-being in the youth.

The UPRIGHT programme´s conceptual framework is structured in four different domains including skills for coping, efficacy, social and emotional learning and mindfulness practice. The intervention was developed by an innovative co-creation process (co-design, co-production and co-customization) participating five European regions representative of the cultural and socioeconomic variability (Lower Silesian in Poland, Basque Country in Spain, Trento in Italy, Denmark and Reykjavik capitol area in Iceland).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents from 1st grade (12-14 years of age) studying in the participating schools, their families and teachers of these adolescents.

Exclusion Criteria:

* None

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4460 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mental well-being | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  The mental well-being is measured by the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS-14) scale in adolescents, families and teachers. This is a 14-item scale with 5 response categories.
Change in resilience capacities for adolescents | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  The resilience is measured by the Resilience Scale for Adolescents (READ-28) for adolescents and designed as a 28-items scale with 5 response categories.

SECONDARY OUTCOMES:
Change in resilience capacities for adults | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  The resilience is measured by the Resilience Scale for adults (RSA-33) for adults and designed as a 33-items scale with 5 response categories
Change in school resilience capacities | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  The school resilience is measured by an ad hoc created scale which was validated under the UPRIGHT project setting.
Change in perceived stress | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  The Perceived Stress Scale (PSS-4) scale is a 4-items tool with 5 response categories (never, almost never, sometimes, fairly often; very often)
Change in the quality of life of adolescents | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  Kidscreen-10 is a 10-items scale with a 5-response options (not at all; slightly; moderately; very extremely)
Change in the cases of bullying, substance use, violence and injuries | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  This outcome is measured by a sub-scale of the Health Behaviour in School-Aged Children (HBSC) including 14-items with 5-response categories
Change in the incidence of anxiety | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  Anxiety is measured by the General Anxiety Disorder (GAD-7)
Change in the incidence of depression | 1st wave: Month 9 (baseline), Month 18 and Month 30. 2nd wave: Month 21 (baseline), Month 30 and Month 42.
  Depression is measured by the Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Carlota Las Hayas, Principal Investigator — Biosistemak Institute for Health Systems Research
Locations (5):
- Aarhus University, Aarhus C, Denmark
- University of Iceland, Reykjavik, Iceland
- Fondazione Bruno Kessler, Trento, Trentino-Alto Adige, Italy
- Urzad Marszalkowski Wojewodztwa Dolnoslaskiego, Wroclaw, Low Silesia, Poland
- Kronikgune, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kieling C, Baker-Henningham H, Belfer M, Conti G, Ertem I, Omigbodun O, Rohde LA, Srinath S, Ulkuer N, Rahman A. Child and adolescent mental health worldwide: evidence for action. Lancet. 2011 Oct 22;378(9801):1515-25. doi: 10.1016/S0140-6736(11)60827-1. Epub 2011 Oct 16. PMID 22008427
- [Background] Pina-Camacho L, Del Rey-Mejias A, Janssen J, Bioque M, Gonzalez-Pinto A, Arango C, Lobo A, Sarro S, Desco M, Sanjuan J, Lacalle-Aurioles M, Cuesta MJ, Saiz-Ruiz J, Bernardo M, Parellada M; PEPs Group. Age at First Episode Modulates Diagnosis-Related Structural Brain Abnormalities in Psychosis. Schizophr Bull. 2016 Mar;42(2):344-57. doi: 10.1093/schbul/sbv128. Epub 2015 Sep 14. PMID 26371339
- [Background] Wathen CN, MacGregor JC, Hammerton J, Coben JH, Herrman H, Stewart DE, MacMillan HL; PreVAiL Research Network. Priorities for research in child maltreatment, intimate partner violence and resilience to violence exposures: results of an international Delphi consensus development process. BMC Public Health. 2012 Aug 21;12:684. doi: 10.1186/1471-2458-12-684. PMID 22908894
- [Background] Masten AS. Ordinary magic. Resilience processes in development. Am Psychol. 2001 Mar;56(3):227-38. doi: 10.1037//0003-066x.56.3.227. PMID 11315249
- [Background] Patel V, Goodman A. Researching protective and promotive factors in mental health. Int J Epidemiol. 2007 Aug;36(4):703-7. doi: 10.1093/ije/dym147. Epub 2007 Jul 23. No abstract available. PMID 17646185
- [Background] Dray J, Bowman J, Campbell E, Freund M, Hodder R, Wolfenden L, Richards J, Leane C, Green S, Lecathelinais C, Oldmeadow C, Attia J, Gillham K, Wiggers J. Effectiveness of a pragmatic school-based universal intervention targeting student resilience protective factors in reducing mental health problems in adolescents. J Adolesc. 2017 Jun;57:74-89. doi: 10.1016/j.adolescence.2017.03.009. Epub 2017 Apr 3. PMID 28384523
- [Derived] Las-Hayas C, Mateo-Abad M, Vergara I, Izco-Basurko I, Gonzalez-Pinto A, Gabrielli S, Mazur I, Hjemdal O, Gudmundsdottir DG, Knoop HH, Olafsdottir AS, Fullaondo A, Gonzalez N, Mar-Medina J, Krzyzanowski D, Morote R, Anyan F, Ledertoug MM, Tidmand L, Arnfjord UB, Kaldalons I, Jonsdottir BJ, de Manuel Keenoy E; UPRIGHT Consortium. Relevance of well-being, resilience, and health-related quality of life to mental health profiles of European adolescents: results from a cross-sectional analysis of the school-based multinational UPRIGHT project. Soc Psychiatry Psychiatr Epidemiol. 2022 Feb;57(2):279-291. doi: 10.1007/s00127-021-02156-z. Epub 2021 Aug 21. PMID 34417859
- [Derived] Las Hayas C, Izco-Basurko I, Fullaondo A, Gabrielli S, Zwiefka A, Hjemdal O, Gudmundsdottir DG, Knoop HH, Olafsdottir AS, Donisi V, Carbone S, Rizzi S, Mazur I, Krolicka-Deregowska A, Morote R, Anyan F, Ledertoug MM, Tange N, Kaldalons I, Jonsdottir BJ, Gonzalez-Pinto A, Vergara I, Gonzalez N, Mar Medina J, de Manuel Keenoy E; UPRIGHT consortium. UPRIGHT, a resilience-based intervention to promote mental well-being in schools: study rationale and methodology for a European randomized controlled trial. BMC Public Health. 2019 Oct 29;19(1):1413. doi: 10.1186/s12889-019-7759-0. PMID 31664974
- See also: Collaborative for academic, social, and emotional learning — https://casel.org/
- See also: Department of Health KidsMatter — https://www.kidsmatter.edu.au/